CLINICAL TRIAL: NCT06921785
Title: A Phase III, Randomised, Open-label, Sponsor-blinded, Multicentre Study of Rilvegostomig in Combination With Bevacizumab With or Without Tremelimumab as First-line Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Phase III Study of Rilvegostomig in Combination With Bevacizumab With or Without Tremelimumab as First-line Treatment of Hepatocellular Carcinoma
Acronym: ARTEMIDE-HCC01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7029C00001
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tremelimumab; Bevacizumab; atezolizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be conducted "Sponsor-blinded", Sponsor personnel directly involved in the study conduct will not have access to efficacy data aggregated by intervention arm prior to study unbinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Tremelimumab , rilvegostomig and bevacizumab
  Interventions: Drug: Tremelimumab; Drug: Rilvegostomig; Drug: Bevacizumab
- Arm B (Experimental): Rilvegostomig, and bevacizumab
  Interventions: Drug: Rilvegostomig; Drug: Bevacizumab
- Arm C (Active Comparator): Atezolizumab, and bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Tremelimumab — IV therapy
  Arms: Arm A
Drug: Rilvegostomig — IV therapy
  Arms: Arm A; Arm B
Drug: Bevacizumab — IV therapy
Drug: Atezolizumab — IV therapy
  Arms: Arm C

SUMMARY:
This is a Phase III, randomised, open-label, sponsor-blinded, 3-arm, multicentre, global study assessing the efficacy and safety of rilvegostomig in combination with bevacizumab with or without tremelimumab compared to atezolizumab in combination with bevacizumab. This study will be conducted in participants with advanced HCC who are not amenable to curative therapy or locoregional therapy

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and tolerability of rilvegostomig in combination with bevacizumab with or without tremelimumab as first-line treatment in participants with advanced HCC. The study comprises 2 parts - a safety lead-in and a randomised period. Prior to the start of the randomised period of the study, a single-arm safety lead-in period will be applied to evaluate the safety and tolerability of rilvegostomig in combination with bevacizumab and tremelimumab.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable HCC
* WHO/ECOG performance status of 0 or 1
* BCLC stage B (that is not eligible for locoregional therapy) or stage C. Child-Pugh Score class A
* At least one measurable target lesion
* co-infected with HBV and HCV are not eligible
* Adequate organ and bone marrow function measured during the screening period
* Must not have received prior systemic therapy for intermediate, advanced, or metastatic HCC.
* Disease that is not amenable to curative surgical and/or locoregional therapies. For participants who received locoregional therapy for HCC, locoregional therapy must have been completed ≥ 28 days prior to the baseline scan for the current study.

Exclusion Criteria:

Medical condition

* Any evidence of uncontrolled intercurrent diseases
* Active or prior documented autoimmune or inflammatory disorders requiring chronic treatment with steroids or other immunosuppressive treatment
* History of another primary malignancy
* Persistent toxicities caused by previous anti-cancer therapy excluding alopecia, not yet improved to Grade ≤ 1 or baseline.
* Clinically meaningful ascites, pleural effusion, or pericardial effusion requiring non-pharmacologic intervention to maintain symptomatic control within 6 months prior to the first scheduled dose.
* History of active primary immunodeficiency or active infection
* History of hepatic encephalopathy
* Current or recent (within 10 days of first dose of study treatment) use of aspirin (≥ 325 mg/day) or treatment with dipyridamole, ticlopidine, clopidogrel, and cilostazol
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purposes is ineligible

Bleeding or other risks

HCC related

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Central nervous system metastases or spinal cord compression (including asymptomatic and adequately treated disease)
* Prior treatment with anti-CTLA-4 and/or anti-TIGIT.
* Radiotherapy within 28 days and abdominal/ pelvic radiotherapy within 60 days prior to initiation of study treatment, except palliative radiotherapy to bone lesions within 7 days prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2029-03-16 (Estimated); Study Completion 2030-03-14 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the efficacy of Arm A relative to Arm C by assessment of OS in participants with advanced HCC | Up to approximately 6 years
  OS is defined as the time from randomisation until the date of death due to any cause.

SECONDARY OUTCOMES:
To demonstrate the efficacy of Arm B relative to Arm C by assessment of OS in participants with advanced HCC | Up to approximately 6 years
  OS is defined as the time from randomisation until the date of death due to any cause.
To further demonstrate the efficacy of Arm A relative to Arm C and Arm B relateive to Arm C in participants with advanced HCC | Up to approximately 6 years
  PFS according to RECIST 1.1
To further demonstrate the efficacy of Arm A relative to Arm C and Arm B relateive to Arm C in participants with advanced HCC | Up to approximately 6 years
  ORR according to RECIST 1.1
To demonstrate the efficacy of Arm A relative to Arm B in participants with advanced HCC | Up to approximately 6 years
  OS
To demonstrate the efficacy of Arm A relative to Arm B in participants with advanced HCC | Up to approximately 6 years
  PFS
To demonstrate the efficacy of Arm A relative to Arm B in participants with advanced HCC | Up to approximately 6 years
  ORR
To demonstrate the efficacy of Arm A relative to Arm B in participants with advanced HCC | Up to approximately 6 years
  DoR
To demonstrate the efficacy of Arm A relative to Arm C in the population defined by PD-L1 expression subgroups | Up to approximately 6 years
  Association of PD-L1 expression level with:
  • OS
To demonstrate the efficacy of Arm A relative to Arm C in the population defined by PD-L1 expression subgroups | Up to approximately 6 years
  Association of PD-L1 expression level with:
  • PFS per RECIST 1.1
To demonstrate the efficacy of Arm A relative to Arm C in the population defined by PD-L1 expression subgroups | Up to approximately 6 years
  Association of PD-L1 expression level with:
  • ORR per RECIST 1.1
To demonstrate the efficacy of Arm A relative to Arm C in the population defined by PD-L1 expression subgroups | Up to approximately 6 years
  Association of PD-L1 expression level with:
  •DoR per RECIST 1.1
To demonstrate the efficacy of Arm B relative to Arm C in the population defined by PD-L1 expression subgroups | Up to approximately 6 years
  Association of PD-L1 expression level with:
  OS
To demonstrate the efficacy of Arm B relative to Arm C in the population defined by PD-L1 expression subgroups | Up to approximately 6 years
  Association of PD-L1 expression level with:
  PFS per RECIST 1.1
To demonstrate the efficacy of Arm B relative to Arm C in the population defined by PD-L1 expression subgroups | Up to approximately 6 years
  Association of PD-L1 expression level with:
  ORR per RECIST 1.1
To demonstrate the efficacy of Arm B relative to Arm C in the population defined by PD-L1 expression subgroups | Up to approximately 6 years
  Association of PD-L1 expression level with:
  DoR per RECIST 1.1
To investigate the immunogenicity of Arm A and Arm B | Up to approximately 6 years
  Presence of ADAs for tremelimumab and rilvegostomig
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | Up to approximately 6 years
  Occurrence of AEs and SAEs will be graded according to the revised NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (183):
- United States (30):
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Palo Alto, California
  - Research Site, Santa Monica, California
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Fayetteville, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Shreveport, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Blacksburg, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (3):
  - Research Site, Auchenflower
  - Research Site, Camperdown
  - Research Site, Heidelberg
- Brazil (4):
  - Research Site, Porto Alegre
  - Research Site, Santa Maria
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (9):
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (30):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Chongqing
  - Research Site, Deyang
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Hohhot
  - Research Site, Kunming
  - Research Site, Linyi
  - Research Site, Lishui
  - Research Site, Luoyang
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Nantong
  - Research Site, Neijiang
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- France (8):
  - Research Site, Clichy
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Pessac
  - Research Site, Rennes
  - Research Site, Toulouse
- Germany (17):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Moers
  - Research Site, München
  - Research Site, Regensburg
  - Research Site, Ulm
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- India (9):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Binnāguri
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, Vadodara
- Italy (7):
  - Research Site, Bologna
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (28):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Iizuka-shi
  - Research Site, Kashiwa
  - Research Site, Kita-gun
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Mitaka-shi
  - Research Site, Morioka
  - Research Site, Musashino-shi
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Saga
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Suita-shi
  - Research Site, Tokyo
  - Research Site, Toyoake-shi
  - Research Site, Tsu
  - Research Site, Yokohama
- Netherlands (5):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Maastricht
  - Research Site, Rotterdam
  - Research Site, Utrecht
- South Korea (5):
  - Research Site, Busan
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Santander
- Taiwan (7):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Tainan County
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Dusit
  - Research Site, Hat Yai
  - Research Site, Muang
  - Research Site, Ubonratchathani
- Turkey (Türkiye) (5):
  - Research Site, Altındağ
  - Research Site, Ankara
  - Research Site, Erzurum
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (3):
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Manchester
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individualpatient-level data from AstraZeneca group of companies sponsoredclinical trials via the request portal Vivli.org. All requests will be evaluatedas per the AZ disclosure commitment:https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.Yes, indicates that AZ are accepting requests for IPD, but this does notmean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitmentsmade to the EFPIA PhRMA Data Sharing Principles. For details of ourtimelines, please refer to our disclosure commitment athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to theanonymized individual patient-level data via secure research environmentVivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/